CLINICAL TRIAL: NCT00775047
Title: Pharmacist-Administered Injections of Depo-Medroxyprogesterone Acetate for Contraception: A Pilot Randomized Controlled Trial
Brief Title: Pharmacist-Administered Injections for Contraception
Acronym: PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Carla Picardo, MD, MPH, University of North Carolina, Dept. of Social Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-EPID-52
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Contraception
Keywords: depo medroxyprogesterone acetate; Depo Provera; contraceptive compliance; pharmacists; Compliance in receiving additional Depo Provera injections; Satisfaction in receiving Depo Provera injections at a pharmacy compared with usual clinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmacy (Experimental): Women receive their second and third depot-medroxyprogesterone acetate injections at the pharmacy by clinical pharmacists
  Interventions: Other: Pharmacist-administered
- Planned Parenthood clinic (Active Comparator): Women receive their second and third depot-medroxyprogesterone acetate injections per usual care at their Planned Parenthood clinic.
  Interventions: Other: clinic-administered injections

INTERVENTIONS:
Other: Pharmacist-administered — women will receive their injections at a pharmacy by a clinical pharmacist
  Other Names: SQ Depo-Provera
  Arms: Pharmacy
Other: clinic-administered injections — women will return for their injections to the clinic where recruitment took place. They will receive one at 3 months and 6 months.
  Other Names: SQ Depo-Provera
  Arms: Planned Parenthood clinic

SUMMARY:
The purpose of this study is to see if it is a feasible arrangement to have women receive their second and third birth control injection (with Depo-Provera) at a pharmacy compared with receiving it a Planned Parenthood Clinic. Compliance with returning for injections as well as patient satisfaction with the method, providers, and location where injection was received will be assessed and compared between the two sites. The hypothesis is that there will be no difference in return rates for injections at either the pharmacy or the clinic site.

DETAILED DESCRIPTION:
Women who want to use or are currently using Depo-Provera for contraception will be randomized to receive their next two injections either back at the Planned Parenthood clinic or at a local pharmacy where pharmacists are trained to give injections. After each injection, women will be asked to complete a questionnaire to assess their attitudes about the method of birth control, their providers, and the location where they received the injection.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 y.o., English speaking/reading, presenting to Planned Parenthood to use Depo Provera (restarting, first use, or continuing use)

Exclusion Criteria:

* Under 18 years of age, English illiterate (reading and verbal)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2007-09 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Compliance in returning for 3 month and 6 month injections | 3 months and 6 months after first injection

SECONDARY OUTCOMES:
Attitudes about clinical setting | 3 months and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carla Picardo, MD, MPH, Principal Investigator — Dept. of Social Medicine, University of North Carolina
Locations (1):
- Planned Parenthood of Central North Carolina, Chapel Hill, North Carolina, United States